CLINICAL TRIAL: NCT01461161
Title: A Single-Dose, Open-Label, Randomized, Food Effect and Blinded, Randomized, Dose Proportionality Study in Healthy Volunteers With Bardoxolone Methyl
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 402-C-1004
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — bardoxolone methyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 20 mg bardoxolone methyl (Experimental)
  Interventions: Drug: bardoxolone methyl
- 60 mg bardoxolone methyl (Experimental)
  Interventions: Drug: bardoxolone methyl
- 80 mg bardoxolone methyl (Experimental)
  Interventions: Drug: bardoxolone methyl

INTERVENTIONS:
Drug: bardoxolone methyl — oral, single dose

SUMMARY:
This study is to determine the effect of food on a single dose of 20 mg bardoxolone methyl administered to normal healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females between 18 and 45 years of age;
2. Willing to practice methods of birth control (both males who have partners of childbearing potential and females of childbearing potential) during screening, while taking study drug and for at least 30 days after the last dose of study drug is ingested;
3. Female subjects of childbearing potential must be non-pregnant and non-lactating and have a negative serum pregnancy test result prior to enrollment into the trial;
4. Body mass index (BMI) between 19 and 31 kg/m2;
5. Willing and able to give written informed consent for study participation and provide consent for access to medical data according to appropriate local data protection legislation, allowing authorization to access medical records that describe events captured in the endpoints;
6. Willing and able to cooperate with all aspects of the protocol.

Exclusion Criteria:

1. Participated in another clinical trial of an investigational drug (or a medical device) within the last 30 days, or are currently participating in another trial of an investigational drug (or a medical device);
2. Any condition possibly affecting absorption, distribution, metabolism or excretion of drugs that may confound the analyses conducted in this study [e.g., previous surgery on the gastrointestinal tract that includes removal of parts of stomach, bowel, liver, gall bladder, or pancreas];
3. Known hypersensitivity to any component in the formulation of the study drug, bardoxolone methyl;
4. Evidence or history of or concurrent clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dose administration), hematological, endocrine, immunological, renal, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease that in the judgment of the investigator could potentially either pose a health risk to the subject during the study or influence the study outcome;
5. Evidence of hepatic or biliary dysfunction including elevation of total bilirubin, direct bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), gamma glutamyl transpeptidase (GGT), lactate dehydrogenase (LDH), or alkaline phosphatase levels to greater than the upper limit of normal (ULN);
6. Positive test results for human immunodeficiency virus type 1 or 2 antibody, hepatitis B surface antigen, or hepatitis C virus antibody at screening;
7. Any medical or dental procedure, no matter how minor, that is planned or anticipated to occur during the conduct of the study;
8. History of drug or alcohol abuse or dependence within the last year;
9. Any vaccination within 30 days before start of this study and throughout the study;
10. Use of or need for any systemic drug(s) including vitamins or herbal preparations other than drugs used for contraception, within 30 days before entry into the study or during the study;
11. Use of aspirin, non-steroidal anti-inflammatory agents, or acetaminophen within 5 days prior to the ingestion of the study drug; use of aspirin or non-steroidal anti inflammatory agents (but not acetaminophen) will be allowed for isolated episodes of pain at the discretion of the investigator;
12. Donation or receipt of blood or blood components within the 4 weeks prior to the study. The investigator should instruct subjects who participate in this study not to donate blood or blood components for 4 weeks after the completion of the study;
13. Any diagnostic or intervention procedure requiring a contrast agent within the 30 days prior to study participation;
14. Sustained systolic blood pressure > 140 mmHg or < 100 mmHg or a diastolic blood pressure > 95 mmHg at screening or baseline measured after 5 minutes in a sitting position. Blood pressure may be re-tested twice in a sitting position at intervals of 5 minutes. The pressure elevation is considered sustained if either the systolic or the diastolic pressure exceeds the stated limits after three assessments;
15. A pulse rate at rest of < 45 bpm or > 100 bpm;
16. Abnormal screening ECG which is interpreted by the investigator to be clinically significant;
17. Used tobacco-containing products (e.g., cigarettes, cigars, chewing tobacco, snuff, etc.) or products for smoking cessation 2 weeks prior to Day -1 of Period 1 of the study;
18. Consumed alcohol or xanthine-containing products (e.g., tea, coffee, chocolate, cola, etc.) within 72 hours prior to Day -1 of Period 1 of the study;
19. Treated within 30 days before Day -1 of Period 1, 5 half-lives or twice the duration of biological effect of the previous investigational drug (whichever is longer) with any investigational agent;
20. A positive history of drug abuse or who test positive for drug(s) of abuse, ethanol, amphetamines, barbiturates, cocaine, opiates, benzodiazepines, cannabinoids or cotinine (indicating active current smoking) at the screening or Day -1 of Period 1 visit;
21. Female subjects who are planning a pregnancy or are pregnant or lactating;
22. Deemed by the investigator to be inappropriate for this study, including subjects who are unable to communicate with the investigator due to language problems, poor mental development, or impaired cerebral function;
23. Any concurrent clinical conditions that in the judgment of the investigator could either potentially pose a health risk to the subject while involved in the study or could potentially influence the study outcome.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2011-10-31 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

PRIMARY OUTCOMES:
Effect of food on Pharmacokinetics of a 20 mg single dose of bardoxolone methyl | 28 Days

SECONDARY OUTCOMES:
Dose proportionality of 20mg, 60mg, and 80mg bardoxolone methyl | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical Research, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/